CLINICAL TRIAL: NCT05423665
Title: Speckle Tracking Echocardiography as a Tool for Early Diagnosis of Impaired Fetal Growth in Twin Pregnancies
Brief Title: Speckle Tracking Echocardiography as a Tool for Early Diagnosis of Impaired Fetal Growth Twin Pregnancies
Acronym: HEART
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other); Maxima Medical Center (Other); Hasselt University (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0193
Record Dates: First submitted 2022-05-31; First posted 2022-06-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Fetal Growth Restriction; Cardiac Remodeling, Ventricular; Placental Insufficiency; Air Pollution
MeSH Terms: conditions — Fetal Growth Retardation; Ventricular Remodeling; Placental Insufficiency | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal growth restricted: Observation of cardiac remodeling perinatal and postnatal
  Interventions: Other: sample collection
- Appropriately grown: Observation of cardiac remodeling perinatal and postnatal
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — blood sample at 21 weeks of gestation clips of the fetal heart at 21 weeks of gestation, 30 weeks of gestation and 1-3 days after birth collection of umbilical cord blood at birth collection of the placenta at birth

SUMMARY:
In this project there are 2 time points during the pregnancy included, namely at 21 weeks and 30 weeks of gestation, to measure the predictive values of FGR, strain and strain rate. The fetal growth parameters will be collected at the same time points, to define the growth (differences) throughout gestation of both fetuses. A maternal blood sample will be taken at 21 weeks of gestation to identify the level of exposure to air pollution (black carbon) and the level of biochemical markers of placental dysfunction. Doppler ultrasounds will be used for antenatal identification of placenta insufficiency. At birth, umbilical cord blood and the placenta will be collected. The placenta will be examined, to identify morphological findings which are associated with FGR. The umbilical cord blood and placental biopsy will be used for the level of exposure to air pollution and the level of oxidative stress. One to three days after birth, neonatal strain and strain rate will be measured to define postnatal cardiac remodeling as well as the neonatal blood pressure as cardiovascular risk factor.

DETAILED DESCRIPTION:
Fetal growth restriction (FGR) is diagnosed in 5-10% of the pregnancies. After preterm birth, it is the second leading cause of perinatal morbidity and mortality. Twin pregnancies have a higher occurrence of FGR than singletons, in monochorionic (MC) twin pregnancies it's diagnosed in 19.7% of the cases and in dichorionic (DC) twin pregnancies in 10.5% of the cases. Fetuses with FGR are at greater risk of perinatal morbidity and mortality and even long-term health defects. From a public health perspective, it's important to correctly diagnose FGR to adjust the antenatal and postnatal care and to have more insight into the factors influencing early onset cardiovascular disease. STE has a strong predictive value for cardiovascular function, therefore it would be a promising tool to add in the routine pregnancy clinical care. Speckle tracking echocardiography (STE) is a relative new technique especially in the pregnancy follow up, which permits offline calculation of myocardial velocities and deformation parameters. These parameters, including strain and strain rate, provide information about the fetal myocardial function. Apart from investigating if STE can be used for the prediction of FGR, we will also investigate the association between fetal exposure to air pollution and in utero cardiac remodeling. Indeed, it is known that inhalation of particulate matter (e.g. black carbon) during the pregnancy can reach the placenta and lead to alterations in the placenta's function including increases in oxidative stress markers. Early life exposure to black carbon has been associated with adverse cardiovascular health outcomes and reduction of fetal growth, especially in multiple gestation pregnancies.

In this project we will include 2 time points during the pregnancy, namely at 21 weeks and 30 weeks of gestation, to measure the predictive values of FGR, strain and strain rate. The fetal growth parameters will be collected at the same time points, to define the growth (differences) throughout gestation of both fetuses. A maternal blood sample will be taken at 20 weeks of gestation to identify the level of exposure to air pollution (black carbon) and the level of biochemical markers of placental dysfunction. Doppler ultrasounds will be used for antenatal identification of placenta insufficiency. At birth, umbilical cord blood and the placenta will be collected. The placenta will be examined, to identify morphological findings which are associated with FGR. The umbilical cord blood and placental biopsy will be used for the level of exposure to air pollution and the level of oxidative stress. One to three days after birth, neonatal strain and strain rate will be measured to define postnatal cardiac remodeling as well as the neonatal blood pressure as cardiovascular risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or dichorionic twin pregnancy
* Pregnant women 21 weeks ( ± 2 weeks) of gestation at the first visit
* Women ≥ 18 years

Exclusion Criteria:

* Women pregnant of multiples of higher order (≥3 siblings) Monochorionic twin pregnancy
* Fetal arrhythmia
* Known fetal congenital or genetic abnormalities
* Any suspicion of congenital fetal anomalies that might influence fetal cardiac function
* Pre-existing maternal hypertensive disease
* Autoimmune disease including systemic lupus erythematosus
* History of stillbirth
* Diabetes mellitus (mother)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: The number of subjects that will be included in this study is: 600 neonates (200 twin pairs and 200 singletons) and 400 pregnant mothers.
  The fetuses are divided into following sub-groups:
  * Appropriately grown
  * Fetal growth restricted
  * Selective fetal growth restricted (specific for twins)
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
To assess the change in strain measured by speckle tracking echocardiography as a tool for early diagnosis of impaired fetal growth in multiple gestations | Prenatal to 1-3 days after birth
  to determine the change in fetal strain and strain rate in twin pregnancies in comparison with fetal growth
To determine the intra-pair differences in fetal growth and strain (cardiac remodeling) in multiple gestations. | Prenatal to 1-3 days after birth
  to compare changes in strain and strain rate with fetal growth within 1 twin pair
To compare the strain values (cardiac remodeling) between singletons and twin pregnancies | Prenatal to 1-3 days after birth
  to compare the changes in strain and strain rate between singletons and twin pregnancies

SECONDARY OUTCOMES:
To investigate the association between placenta functioning and in utero cardiac remodeling | Prenatal to 1-3 days after birth
  to evaluate placenta insufficiency (Doppler ultrasound, biochemical marker) with strain and strain rate
To explore in utero cardiac remodeling in association with neonatal cardiovascular health | Prenatal to 1-3 days after birth
  to evaluate strain and strain rate with the neonatale blood pressure and heart rate
To study the association between prenatal air pollution exposure and in utero cardiac remodeling | Prenatal to 1-3 days after birth
  to evaluate prenatal air pollution (black carbon particles in blood sample mother and placenta) with strain and strain rate
To investigate placenta functioning as a mediator between air pollution and cardiac remodeling | Prenatal to 1-3 days after birth
  To evaluate prenatal air pollution (black carbon particles in blood sample mother and placenta) with placenta insufficiency (biochemical marker, Doppler ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Kristien Roelens, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - Universitair ziekenhuis Leuven, Leuven
- Maxima medical center, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided